CLINICAL TRIAL: NCT04935346
Title: Awareness of Dysphagia in Medical and Nursing Students
Brief Title: Dysphagia Awareness In Medical and Nursing Students
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPMRTRHadimns
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Dysphagia; Awareness; Students
Keywords: dysphagia; awareness; medical students; nursing students
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention group — The awareness of medical and nursing students were evaluated. there is no intervention

SUMMARY:
A survey consisting of questions about swallowing and dysphagia was provided to universities' medicine and nursing students. The answers of students were analyzed

DETAILED DESCRIPTION:
The undergraduate training of health care professionals may provide the necessary theoretical and practical approach to future nurses and physicians. This study was planned to investigate students' dysphagia knowledge level and awareness in the medicine and nursing faculties. A survey consisting of questions about swallowing and dysphagia was provided to universities' medicine and nursing students. The answers of students were analyzed

ELIGIBILITY:
Inclusion Criteria:

* The fourth, fifth, and sixth-grade students in the faculty of medicine
* The second, third, and fourth-grade students in the nursing faculty

Exclusion Criteria:

* The first, second and third-grade students in the faculty of medicine
* The first grade students in the nursing faculty

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was conducted with students at medical and nursing faculties in Turkey
Sampling Method: Probability Sample
Enrollment: 1203 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
A survey | Participants completed the survey at once. 20 minutes required to complete the survey
  A survey that consists of questions related to dysphagia awareness

CONTACTS AND LOCATIONS:
Overall Officials: Betül Yavuz Keleş, MD, Principal Investigator — Istanbul physical Medicine and Rehabilitation Training and Research Hospital; Sibel Eyigör, prof, Study Director — Ege University
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and research Hospital, Istanbul, Turkey (Türkiye)